CLINICAL TRIAL: NCT07001618
Title: A Randomized Multicenter Phase II Trial Evaluating Oral Pooled Fecal Microbiotherapy (MaaT033) Concomitant to Cemiplimab (CB) Versus Best Investigator's Choice (BIC) in Resistance to PD-1/PD-L1 Blockade Due to Antibiotics (ATB) Uptake in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Oral Pooled Fecal Microbiotherapy (MaaT033) Concomitant to Cemiplimab Versus Best Investigator's Choice in Patients With Resistance to Treatment Due to Antibiotics Uptake With Advanced Non-small Cell Lung Cancer
Acronym: IMMUNOLIFE2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: MaaT Pharma (Industry); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-517018-14-00; 2024/3967 (Other: CSET Number (Gustave Roussy ID))
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: MAAT033; ORAL POOLED FECAL MICROBIOTHERAPY; ADVANCED NON SMALL CELL LUNG CANCER; ANTIBIOTICS INDUCED RESISTANCE
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab; Cisplatin; Carboplatin; Pemetrexed; Bevacizumab; Paclitaxel; Gemcitabine; Docetaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination of MaaT033 + Cemiplimab (CB) (Experimental): CB will be administered every 3 weeks. Oral pooled fecal microbiotherapy MaaT033 will be taken by patient (capsules) for a week before CB administration, repeated every other 3 weeks for 6 months.
  Interventions: Drug: MaaT033 capsule; Drug: Cemiplimab
- Best Investigator's Choice (BIC) (Active Comparator): Patients will receive chemotherapy according to current standard of care protocols according to investigator's best choice from current guidelines combinations.
  Interventions: Drug: Cisplatin; Drug: Carboplatine; Drug: Pemetrexed (Alimta); Drug: Bevacizumab; Drug: Paclitaxel; Drug: gemcitabine; Drug: Docetaxel; Drug: Vinorelbine i.v. 25 mg/m²; Drug: Vinorelbine oral

INTERVENTIONS:
Drug: MaaT033 capsule — MaaT033 capsule will be taken orally once a day for a week before every Cemiplimab cycle for the first 6 months of treatment.
  Arms: Combination of MaaT033 + Cemiplimab (CB)
Drug: Cemiplimab — CB will be administered 350 mg IV over 30 minutes every 21 days up to 2 years
  Other Names: LIBTAYO
  Arms: Combination of MaaT033 + Cemiplimab (CB)
Drug: Cisplatin — 75mg/m2 at day 1 (d1) every 21 days (q21)
  Arms: Best Investigator's Choice (BIC)
Drug: Carboplatine — Area Under the Curve (AUC) 5-6 at d1 q21
  Arms: Best Investigator's Choice (BIC)
Drug: Pemetrexed (Alimta) — 500mg/m2 at day 1 (d1) q21
  Arms: Best Investigator's Choice (BIC)
Drug: Bevacizumab — 10mg/kg at d1 and day 15 (d15) every 28 days (q28)
  Arms: Best Investigator's Choice (BIC)
Drug: Paclitaxel — 175mg/m2 at d1 q21 or 80 mg/m2 at d1, day 8 (d8), day 15 q28
  Arms: Best Investigator's Choice (BIC)
Drug: gemcitabine — 1250 or 1000 mg/m2 d1, d8 q21
  Arms: Best Investigator's Choice (BIC)
Drug: Docetaxel — 75 mg/m2 d1 q21 or 33mg/mq d1, d8 q21 q21
  Arms: Best Investigator's Choice (BIC)
Drug: Vinorelbine i.v. 25 mg/m² — 25-30 mg/m2 d1, d8 q21
  Arms: Best Investigator's Choice (BIC)
Drug: Vinorelbine oral — 30 mg/50 mg per os 3 days per week (metronomic)
  Arms: Best Investigator's Choice (BIC)

SUMMARY:
The goal of IMMUNOLIFE2 is to overcome primary resistance to immune checkpoint inhibitors (ICIs), such as pembrolizumab or nivolumab used alone or in combination with chemotherapy, observed in patients with advanced non-small cell lung cancer (NSCLC) following antibiotic exposure, which induces intestinal dysbiosis. The reintroduction of immunotherapy with Cemiplimab, combined with oral pooled fecal microbiotherapy (MaaT033), aims to restore gut microbiota and potentially reverse resistance to ICIs.

The main objective is to determine whether the combination of MaaT033 and Cemiplimab provides a superior disease control rate compared to the current best investigator's choice as comparator.

Patients will be randomized to receive either:

* Experimental arm: MaaT033 administered orally for one week prior to each cycle of Cemiplimab, which will be given in hospital care every 3 weeks for 6 months, followed by Cemiplimab alone thereafter;
* Control arm: Best investigator's choice

DETAILED DESCRIPTION:
IMMUNOLIFE2 is a randomized Phase II clinical trial multicenter aiming at circumventing primary resistance to ICI observed in patients with advanced NSCLC following ATB uptake in the harmful window using FMT strategy (oral pooled fecal microbiotherapy MaaT033) concomitant to CB. Hence the IMMUNOLIFE2 trial described here is exploring the possibility of an improvement of DCR to CB in patients with ICI resistance due to ATB-induced gut dysbiosis. This will be an outstanding opportunity to explore a therapeutic strategy to surpass ATB mediated resistance but for any cause of intestinal dysbiosis that compromise anti-PD1-based therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are at least 18 years of age on the day of signing informed consent,
2. All participants must understand spoken and written national language,
3. Histologically confirmed diagnosis of NSCLC (adenocarcinoma versus squamous cell carcinoma versus others)
4. Have metastatic or unresectable NSCLC and considered by their physician to be indicated for a new line of immunotherapy.
5. Have an Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 to 2. Evaluation of ECOG-PS is to be performed within 7 days prior to the date of treatment allocation.
6. Patients who have progressed after immunotherapy or immunotherapy plus platinum-based chemotherapy (with platinum-based chemotherapy and ICI either sequentially or concomitantly).
7. Have received ATB within 60 days before and 42 days after the first ICI administration and have progressed within 6 months after the first ICI.
8. There are no restrictions on the number of prior lines of treatment. Patients may be included regardless of the number of previous therapies received.
9. A male participant must abstain from heterosexual activity or must agree to use a contraception as detailed below (or in Appendix 2 of this protocol) during the treatment period and for at least 9 months after the last dose of CB or BIC and refrain from donating sperm during this period. (In application of the new recommendations of the CTFG)
10. A female participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and if at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2.
    2. A WOCBP should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. A WOCBP must agree to follow the contraceptive guidance in Appendix 2 or abstain from heterosexual activity during the treatment period and for at least 180 days, after the last dose of treatment.
11. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
12. Patients must be affiliated to a social security system or beneficiary of the same
13. Have an estimated life expectancy greater than 3 months (from inclusion).
14. Meet acceptable steroid dose thresholds (i.e., not above the acceptable threshold <10 mg prednisone daily or equivalent) if receiving systemic steroids at physiologic doses
15. Have measurable disease based on RECIST 1.1 criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
16. Have adequate organ function as defined in the Table 1. All screening laboratory tests must be performed within 28 days prior to the start of study treatment.

Exclusion Criteria:

1. Immunodeficiency or systemic steroid therapy equivalent to prednisolone >10mg/day or equivalent within 7 days prior to the first dose of trial treatment.
2. Active ongoing infection requiring ATB treatment.
3. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years prior to enrollment. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Participants who have entered the follow-up phase of an investigational study may participate if it has been 4 weeks after the last dose of the previous investigational agent and that all study drug-related AEs have resolved to grade 1 or less.
7. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has a known history of Human Immunodeficiency Virus (HIV).
10. Has a known history of Hepatitis B virus (HBV, defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (HCV, considered active if HCV RNA is detected) infection. Note: no testing for HBV and HCV is required unless mandated by local health authority.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Any condition which, in the Investigator's opinion, makes it undesirable for the subject to participate in a clinical trial or which would jeopardize compliance with the protocol.
13. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
14. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of treatment.
15. Persistent toxicities related to prior treatment of grade greater than 1.
16. Swallowing disorders which can affect the intake of the oral pooled fecal microbiotherapy (MaaT033).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | At 12 weeks and confirmation 4-8 weeks from the initial response assessment.
  Percentage of patients who have not shown disease progression regarding complete response, partial response, stable disease as per RECIST 1.1 criteria.
  Confirmation of response must be demonstrated with an assessment 4-8 weeks from the initial response assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At 12 months, 24 months, 36 months and 60 months.
  Percentage of patients who have not shown disease progression regarding complete response and partial response as per RECIST 1.1 criteria.
Progression free survival (PFS) | At 12 months, 24 months, 36 months and 60 months.
  The PFS is defined as the time from random assignment to the progression, or death due to any cause, whichever occurs first.
Overall survival (OS) | At 12 months, 24 months, 36 months and 60 months.
  The OS is defined as the time from random assignment to the date of death due to any cause, or to the date of censoring at the last time the subject was known to be alive.
Duration of response | At 12 months, 24 months, 36 months and 60 months.
  The DoR is defined as the time from the first confirmed patient response (CR or PR) to disease progression (or death from any cause).
Incidence of AEs | At end of study, 60 months.
  Incidence of AEs will be summarized using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0. Safety parameters include all SAEs or non-serious adverse events (AEs) and deaths graded using the NCI-CTCAE v5.0 (Common Terminology Criteria for AEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: No